CLINICAL TRIAL: NCT02503410
Title: Augmenting Back Pain Exercise Therapy Using an Interactive Gaming-based Intervention in the Home Setting
Brief Title: An Interactive Gaming-based Intervention for Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding to continue the study
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, PhD, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-P-000663
Record Dates: First submitted 2015-07-10; First posted 2015-07-21 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: lower back; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor is blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Active Comparator): Subjects receive physical therapy for low back pain as typically prescribed in the clinic.
  Interventions: Behavioral: Usual care
- Interactive gaming (Experimental): Subjects participate in an intervention combining usual care and home-based exercises using the Valedo system.
  Interventions: Behavioral: Interactive gaming

INTERVENTIONS:
Behavioral: Usual care — Subjects receive standard physical therapy, including outpatient visits as prescribed by the treating clinician and home-based exercises based on recommendations by the physical therapist.
  Arms: Usual care
Behavioral: Interactive gaming — Subjects receive a combination of standard physical therapy in the clinic and home-based exercises that they perform using the Valedo system.
  Arms: Interactive gaming

SUMMARY:
This study aims to compare the outcomes of a traditional, exercise-based rehabilitation intervention for chronic low back pain with the outcomes achieved by combining a traditional intervention with adjunct therapy delivered using an interactive gaming-based system for home-based therapy.

DETAILED DESCRIPTION:
The study relies upon the Valedo system by Hocoma AG to implement an interactive gaming-based intervention (i.e. subjects receive part of their physical therapy by playing interactive video games). The system is similar to consumer electronics products for interactive gaming that track the subject's movements using body-worn sensors. The FDA has determined that the Valedo system is a 510(K) exempt device under the product code ION (i.e. exerciser, non-measuring device for Physical Medicine). In the study, subjects with non-specific chronic low back pain are randomized using a block design to one of two groups: group 1 receives usual care alone; group 2 receives an exercise-based rehabilitation intervention using interactive gaming in addition to usual care. Clinical assessments are performed at baseline and again 4 weeks and 8 weeks after baseline measures are gathered.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Back pain subject-rated > 3 on an 11 point visual-analog scale (0-10), with pain reported for a time > 6 months
* Able to commit to all study visits
* Low back pain attributable to mechanical etiology as opposed to infectious, neoplastic, or inflammatory causes.
* BMI ≤ 40
* Familiar with tablet use

Exclusion Criteria:

* Vision or mobility impairment interfering with the performance of the interactive games
* Current or anticipated receipt of payments from Worker's Compensation or other insurance for disability attributed to low back pain
* Additional treatment for back pain during the period of the study, such as acupuncture
* Unresolved musculoskeletal pathology of the lower limbs
* Severe radiculopathic pain
* Alcohol or substance abuse
* Prior discectomy or implantation of rods, screws or plates (bulging disc without radicular pain is not exclusionary; hip or shoulder replacement is not exclusionary)
* Current medication with coumadin or prednisone, chronic use of steroid medications, daily use of narcotic analgesics, or estrogen supplementation, tricyclic anti-depressants (if not on a regular steady dose at least one month prior to enrollment), or any substance that could impair balance.
* Current diagnosis of:

  1. Balance problems due to vestibular or other neurological impairments.
  2. Osteoporosis (Osteopenia is not an exclusionary condition)
  3. Fibromyalgia
  4. Severe or progressive neurological deficits, including neuromotor impairment
  5. Any hypercoagulation condition
  6. Eczema, Psoriasis, or skin infections, and deep vein thrombosis
  7. Burns or other acute trauma including unhealed bone fractures or open wounds
  8. Psychiatric illness not well controlled, or current episode of exacerbated major depressive disorder
  9. Rheumatoid arthritis
* Any other major medical condition that would impair the subject's ability to complete the study visits
* Any other major medical condition that has not been stabilized, or that would impair the subject's ability to complete the activities required by the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited primarily among the outpatient population of individuals with low back pain at Spaulding Rehabilitation Hospital.
Period: Overall Study
Arm/Group | Usual Care | Interactive Gaming
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Interactive Gaming | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.4) | 31.7 (3.8) | 34.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7
Visual Analog Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Subjects are asked to indicate their pain level using a visual analog scale, namely they are asked to choose the position on a horizontal line - drawn on a piece of paper - that corresponds to the pain level that they experience. The line is about 10 cm long and is divided into 10 intervals of equal length referred to as units. The minimum value on the scale is zero (meaning no pain). The maximum value on the scale is ten (meaning maximum ever experienced pain).
  units on a scale | 3.5 (1.3) | 4.0 (1.0) | 3.7 (1.1)
Pain Frequency [Mean (Standard Deviation); unit: days] — Subjects are asked how many days they experienced low back pain during the week prior to the study visit.
  days | 5.3 (0.9) | 6.0 (1.7) | 5.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Pain Scale at 4 Weeks
Description: Subjects are asked to indicate their pain level using a visual analog scale, namely they are asked to choose the position on a horizontal line - drawn on a piece of paper - that corresponds to the pain level that they experience. The line is about 10 cm long and is divided into 10 intervals of equal length referred to as units. The minimum value on the scale is zero (meaning no pain). The maximum value on the scale is ten (meaning maximum ever experienced pain).
Time Frame: Change from baseline in Visual Analogue Pain Scale score at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care Group: physical therapy (as prescribed during 8 to 12 weeks) and home exercises (at least 2x/week)
  Home-based exercises: Subjects will receive a combination of physical therapy and home exercise program during 8 to 12 weeks. Home exercise will be recommended at least two times a week. Usual Care of LBP provided in SRH consists of exercises and manual therapy in various combinations according to the needs of the subject. Subjects will fill out a questionnaire about their pain and how much time they spent doing the home exercises every two weeks.
- Interactive Home-Based System Group: physical therapy (as prescribed during 8 to 12 weeks) and interactive exercises program at home with the Valedo® System (Hocoma AG) (at least 2x/week)
  Interactive gaming home-based exercises: Subjects will receive a combination of physical therapy (during 8 to 12 weeks) and at least two sessions of interactive exercises program at home with the Valedo® System (Hocoma AG). Subjects will fill out a questionnaire about their pain every two weeks during the treatment period.
  Valedo® System (Hocoma AG)
Arm/Group | Usual Care Group | Interactive Home-Based System Group
Number analyzed (Participants) | 4 | 3
units on a scale | 0.0 (0.8) | 0.3 (1.2)

2. Primary Outcome: Visual Analogue Pain Scale at 8 Weeks
Description: as for outcome 1
Time Frame: Change from baseline in VAS score at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
units on a scale | 0.2 (1.7) | 1.3 (1.2)

3. Primary Outcome: Pain Frequency at 4 Weeks
Description: Subjects are asked how many days they experienced low back pain during the week prior to the study visit.
Time Frame: Change in pain frequency at 4 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
days | 2.5 (2.4) | -0.3 (0.6)

4. Primary Outcome: Pain Frequency at 8 Weeks
Description: Subjects are asked how many days they experienced low back pain during the week prior to the study visit.
Time Frame: Change in pain frequency at 8 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
days | -0.2 (2.1) | 0.0 (0.0)

5. Secondary Outcome: Oswestry Low Back Pain Disability Questionnaire at 4 Weeks
Description: Subjects are asked to fill in a questionnaire inquiring about how their pain interferes with their activities of daily living. Accordingly, they receive a disability score ranging between 0 and 100%. A score between 0 and 20% indicates minimal disability; a score between 21 and 40% indicates moderate disability; a score between 41 and 60% indicates severe disability; a score between 61 and 80% indicates that pain impinges on all aspects of the patient's life; and score between 81 and 100% indicates that the subject is bed-bound.
Time Frame: Change in disability score at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage disability
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
percentage disability | 1.0 (3.5) | 4.7 (4.6)

6. Secondary Outcome: Oswestry Low Back Pain Disability Questionnaire at 8 Weeks
Description: as for outcome 5
Time Frame: Change in disability score at 8 weeks
Measure: Mean (Standard Deviation); unit: percentage disability
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
percentage disability | 12.7 (10.6) | 11.3 (7.0)

7. Secondary Outcome: SF36 at 4 Weeks
Description: The SF36 is a clinical outcome measure based on the administration of a questionnaire inquiring about the quality of life and health status of the subject. It consists of eight normalized (so that they have the some weight) scores related to vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The lower the score the more disability. The higher the score the less disability. The score is provide as units on a scale from 0 to 100.
Time Frame: Change in clinical score at 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
units on a scale | 2.6 (14.6) | 6.6 (11.2)

8. Secondary Outcome: SF36 at 8 Weeks
Description: as for outcome 7
Time Frame: Change in clinical score at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Interactive Gaming
Number analyzed (Participants) | 4 | 3
units on a scale | 13.2 (6.1) | 9.5 (15.7)

ADVERSE EVENTS:
Time Frame: We collected information in regard to potential adverse events during the 8 weeks of the study intervention.
Arm/Group | Usual Care | Interactive Gaming
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT02503410/Prot_SAP_000.pdf